CLINICAL TRIAL: NCT00952731
Title: Pre-surgical Phase IIb Trial of Transdermal 4-Hydroxytamoxifen vs. Oral Tamoxifen in Women With Ductal Carcinoma in Situ of the Breast
Brief Title: 4-Hydroxytamoxifen or Tamoxifen Citrate in Treating Women With Newly Diagnosed Ductal Breast Carcinoma in Situ
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Seema Khan, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NWU07-9-02; NCI-2013-00452 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI 07-9-02 (Other: Northwestern University); NCI-2013-00452 (Registry Identifier: Clinical Trials Reporting Program of NCI); P30CA060553 (NIH); N01CN35157 (NIH)
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Results first posted 2015-07-21 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Ductal Breast Carcinoma in Situ; Estrogen Receptor-positive Breast Cancer
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating | interventions — afimoxifene; Tamoxifen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- oral placebo, afimoxifene (Experimental): 4-hydroxytamoxifen gel 2mg/breast applied daily. Oral placebo taken daily.
  Interventions: Drug: oral placebo; Drug: afimoxifene
- tamoxifen citrate, placebo gel) (Active Comparator): Placebo gel applied to the breasts daily. 20mg oral tamoxifen taken daily (taken as two (2) 10mg capsules).
  Interventions: Drug: tamoxifen citrate; Drug: placebo gel

INTERVENTIONS:
Drug: oral placebo — Oral placebo taken daily for 4-10 weeks.
  Other Names: PLCB
  Arms: oral placebo, afimoxifene
Drug: afimoxifene — 2mg/breast applied daily in the form of a gel for 4-10 weeks.
  Other Names: 4-Hydroxy-Tamoxifen; 4-hydroxytamoxifen
  Arms: oral placebo, afimoxifene
Drug: tamoxifen citrate — 20mg oral tamoxifen taken daily (taken as two (2) 10mg capsules) for 4-10 weeks.
  Other Names: Nolvadex; TAM; tamoxifen; TMX
  Arms: tamoxifen citrate, placebo gel)
Drug: placebo gel — Placebo gel applied to breasts daily for 4-10 weeks.
  Other Names: PLCB
  Arms: tamoxifen citrate, placebo gel)

SUMMARY:
This randomized phase II trial is studying 4-hydroxytamoxifen to see how well it works compared with tamoxifen citrate in treating women with newly diagnosed ductal breast carcinoma in situ. Estrogen can cause the growth of breast cancer cells. Hormone therapy using tamoxifen may fight breast cancer by blocking the use of estrogen by the tumor cells. It is not yet known whether topical tamoxifen causes less damage to normal tissue than systemic tamoxifen in treating patients with ductal carcinoma in situ.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled presurgical trial of 0.228% 4-hydroxy-tamoxifen (4-OHT) gel vs. oral tamoxifen (TAM) 20 mg daily. The study population will consist of 112 pre- and postmenopausal women with any grade DCIS, ER positive, non-palpable DCIS with no evidence of invasion found on diagnostic core needle biopsy (DCNB). In order to accrue a total of 112 participants with DCIS over a period of 22 months, 20 eligible participants total will be screened at the three participating institutions per month with a planned average monthly recruitment of 5 participants total per month. We assume that 22 women (20% of the recruited population, 11 women per arm) will be inevaluable because of the presence of unanticipated invasive disease in the therapeutic surgical excisional (TSE) specimen, or the absence of residual DCIS in the TSE, so that a total of 90 women (45 per arm) will be evaluable for the study endpoints. These estimates are based on numbers from the Lynn Sage Database of NU: over the six-year period 2000-2005, the fraction of women diagnosed with DCIS on core needle biopsy who were found to have no residual DCIS in the TSE was 2.5% and that of women with invasive disease (T1a or greater) in the TSE when the DCNB showed pure DCIS was 13.3%, very similar to the data reported by Bonnett et. al. [56] who found that 13% of pure DCIS lesions seen on DCNB (29/122) were in fact invasive in the TSE. With regard to racial/ethnic groups, 25.6% of the DCIS population at NU were of non-European ancestry (18% African, 4% Hispanic, 3.5% other). WU has higher fractions of African American women with DCIS (24% and 21% respectively).

The participants will be consented following diagnostic core needle biopsy at the time of initial surgical consultation. Baseline assessments include medical history, nipple aspirate fluid (NAF) collection, explanation of gel application, BESS questionnaire (symptom assessment) and blood draw for clinical and research labs including plasma estradiol, progesterone and FSH (rushed), CBC, chemistry profile, liver and renal function tests, Factor VIII, von Willebrand Factor, Factor IX, and total protein S, plasma for insulin-like growth factor (IGF-1) and sex hormone-binding globulin (SHBG), and DNA extraction for assessment of polymorphisms in tamoxifen metabolism genes. At Northwestern plasma and RNA from blood will be collected pre- and post-treatment and will be stored for future proteomic and gene expression fingerprinting

No run-in period is planned. The intervention phase will begin within 5 days following randomization and end on the day prior to surgical resection. The 4-OHT group will apply active gel 2 mg daily to each breast for 4-10 weeks and take oral placebo. The TAM group will take 20 mg TAM orally daily and apply gel placebo. The last dose of study medication will be used on the morning of the day prior to surgery.

Participants will be shipped two 100 ml canisters of 4-OHT or placebo gel plus 130 capsules of tamoxifen or oral placebo at the time of randomization. Participants will take study agents for 4-10 week (minimum). However, if surgery needs to be delayed beyond the 8 week study period for clinical reasons (eg scheduling with plastic surgery) the participant will be sent additional medication by mail to allow continuation of therapy until the day before surgery up to a maximum duration of 10 weeks.

On the day prior to surgery, baseline assessments will be repeated (with the exception of menopausal determination and tamoxifen metabolism gene polymorphisms, but with the addition of blood draw for tamoxifen metabolites and E and Z 4-OHT isomer determination). Under unavoidable circumstances, the end of intervention visit will be allowed on the day of surgery prior to TSE. During the TSE breast adipose tissue from the surgical sample will be snap frozen and stored at -800C for measurement of TAM metabolites. The paraffin block of the DCNB and TSE samples will be acquired by the recruiting institution and 10 sections from each specimen submitted to the NU Pathology Core Facility (NU PCF). The sections will be cut in batches (with pre- and post-samples in the same batch), shipped cold, and processed for immunohistochemistry within a week of sectioning.

Compliance assessment will occur through patient diaries, pill counts and the weighing of returned drug (gel) canisters.

Patients will be assessed for adverse events at the post-surgical visit (approximately 7-14 days after surgery) and by phone at 30 days following the last dose of study agent.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of hormone receptor positive (more than 5% cells staining for ER + and/ or PR +), any grade (using definition of Page and Lagios) ductal carcinoma in situ (DCIS) with or without evidence of microinvasion on diagnostic core needle biopsy within the previous 60 days.
2. Women of age ≥ 18 years. Because no dosing or adverse event data are currently available on the use of 4-hydroxytamoxifen in participants <18 years of age, children are excluded from this study but will be eligible for future pediatric trials, if applicable.
3. ECOG performance status ≥1 (Karnofsky ≥70%)
4. Participants must have normal organ and marrow function as defined below:

   1. Leukocytes≥3,000/uL
   2. Absolute neutrophil count (ANC)≥1,500/uL
   3. Platelets≥100,000/uL
   4. Total bilirubin within normal institutional limits
   5. AST (SGOT)/ALT (SGPT)≤1.5 X institutional ULN
   6. Creatinine within normal institutional limits
5. Women of child-bearing potential must agree to practice barrier birth control, abstinence, or use non-hormonal IUDs from the time that the first pregnancy test is performed throughout the duration of the study and for three months after cessation of study drug. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately.
6. Ability to understand and the willingness to sign a written informed consent document.
7. Ability and willingness to schedule surgical resection of DCIS lesion for 4-10 weeks (28-70 days) following the start of study agent.
8. Willingness to avoid exposing breast skin to natural or artificial sunlight (i.e. tanning beds) for the 4-10 weeks of study agent dosing.

Exclusion Criteria:

1. Prior history of, or at high risk to develop, thromboembolic disease will be excluded.
2. Must not have taken exogenous sex hormones since biopsy diagnosing DCIS and must agree not to use exogenous sex hormones while on study.
3. Must not have taken tamoxifen or other selective estrogen receptor modulators (SERMs) within 2 years prior to entering the study. Women who have discontinued SERM therapy because of thromboembolic or uterine toxicity, will be excluded regardless of duration of use.
4. May not be receiving any other investigational agents.
5. History of allergic reactions attributed to compounds of similar chemical or biologic composition to 4-hydroxytamoxifen or tamoxifen.
6. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
7. Pregnant women are excluded from this study because tamoxifen and 4-hydroxytamoxifen has the potential for teratogenic or abortifacient effects. Women are excluded from enrolling within 3 months of the most recent pregnancy. Women must avoid becoming pregnant in the 3 months following the use of study agent.
8. Women must not have breastfed within three months prior to DCNB. Women who are breast feeding are excluded from entry into this trial because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with tamoxifen or 4-hydroxytamoxifen. Women must agree to forego breastfeeding for three months following the use of study agent.
9. Must not have any dermatologic conditions resulting in skin breakdown in the area of gel application.
10. Must not have a history of previous ipsilateral radiation to the affected breast.
11. Must not have had a breast reduction or augmentation within the 6 months prior to first dose of study agents. Patients who have had breast implants more than 6 months prior to first dose of study agents will be eligible.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-12; Primary Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seema Khan, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between November 2009 and July 2011, subjects were recruited at Northwestern University and Washington University. The original accrual goal was 112, however, the study was halted early due to drug supply issues.
Pre-assignment Details: A total of 31 subjects were registered to the study but only 27 were randomized and began the study. Three participants were deemed ineligible and 1 withdrew consent before randomization.
Groups:
- Treatment Gel + Oral Placebo: 4-hydroxytamoxifen gel 2mg/breast applied daily. Oral placebo taken daily.
  oral placebo: Oral placebo taken daily for 4-10 weeks.
  afimoxifene: 2mg/breast applied daily in the form of a gel for 4-10 weeks.
- Placebo Gel + Oral Treatment: Placebo gel applied to the breasts daily. 20mg oral tamoxifen taken daily (taken as two (2) 10mg capsules).
  tamoxifen citrate: 20mg oral tamoxifen taken daily (taken as two (2) 10mg capsules) for 4-10 weeks.
  placebo gel: Placebo gel applied to breasts daily for 4-10 weeks.
Period: Overall Study
Arm/Group | Treatment Gel + Oral Placebo | Placebo Gel + Oral Treatment
Started | 13 | 14
Randomization | 13 | 14
Treatment & Pre-Surgery | 12 | 14
Surgery | 12 | 14
Follow-up | 12 | 14
Completed | 12 | 14
Not Completed | 1 | 0
Not completed — Drug supply expired | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Gel + Oral Placebo | Placebo Gel + Oral Treatment | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Customized [Number; unit: participants]
  40-49 years | 1 | 2 | 3
  50-59 years | 4 | 7 | 11
  60-69 years | 6 | 4 | 10
  70-79 years | 0 | 1 | 1
  80-89 years | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 7 | 11
  White | 8 | 6 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 13 | 14 | 27
Menopausal status [Number; unit: participants]
  Pre-Menopausal | 4 | 3 | 7
  Post-Menopausal | 9 | 11 | 20

OUTCOME MEASURES:

1. Primary Outcome: Difference Between Ki-67 Labeling Index in Tissue Samples Taken at Baseline and Post-treatment
Description: Ki-67 was measured in matched core and excision tissue samples containing DCIS (Ductal Carcinoma In-Situ) lesions, the core sample was at baseline while the excision sample was at surgery (after approximately 4-10 weeks of treatment).
Time Frame: Baseline and after 4-10 weeks of treatment
Population: 18 total subjects were evaluable for immunohistochemistry marker testing including the Ki-67 labeling index. Of the 26 participants who completed study treatment 2 did not have matching samples available for testing and 6 were excluded because of insufficient DCIS lesion in their samples for testing.
Measure: Mean (Standard Deviation); unit: percentage of 300 DCIS cells
Arm/Group | Treatment Gel + Oral Placebo | Placebo Gel + Oral Treatment
Number analyzed (Participants) | 9 | 9
percentage of 300 DCIS cells | -3.4 (5.0) | -5.1 (5.5)

2. Other Pre Specified Outcome: Compare Concentrations of Tamoxifen and Its Metabolites (4-hydroxytamoxifen, Endoxifen, N-desmethyl Tamoxifen (NDT)) Obtained From Samples on the Day of Surgery
Description: Concentrations of tamoxifen and its metabolites: 4-hydroxytamoxifen, endoxifen, and NDT were measured in breast tissue, blood, and Nipple Aspirate Fluid (NAF) that was collected on the day of surgery.
Time Frame: Day of surgery (after approximately 4-10 weeks)
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Drug Metabolite Levels in the Two Study Groups by CYP2D6 Polymorphism Status
Description: Descriptive statistics and confidence intervals will be provided.
Time Frame: 28-70 days
Reporting Status: Not Posted

4. Other Pre Specified Outcome: 4-OHT Affects Known Tamoxifen-modulated Pathways
Description: Descriptive statistics and confidence intervals will be provided.
Time Frame: 28-70 days
Reporting Status: Not Posted

5. Other Pre Specified Outcome: TAM Metabolite Concentrations and Estrogen Response Markers in Nipple Aspiration Fluid (NAF)
Description: Descriptive statistics and confidence intervals will be provided.
Time Frame: 28-70 days
Reporting Status: Not Posted

6. Secondary Outcome: Difference in Mean Score for Vasomotor Symptoms Including Hot Flashes From Baseline to Time of Surgery
Description: Hot flashes were assessed by the Breast Cancer Prevention Trial Eight Symptom Scale (BESS) questionnaire. This questionnaire measures the incidence of a number of symptoms by asking participants how frequently they experienced them on a scale of 0-4 (0 being Not at All and 4 being Extremely often). BESS questionnaire was administered at baseline and time of surgery. The incidence of vasomotor symptoms (including hot flashes, night sweats, and cold sweats) was measured at baseline (Day 0) and end of treatment prior to surgery (at least 4 weeks later or up to 10 weeks, depending on scheduled surgery date), and changes in the mean score for hot flashes were observed.
Time Frame: Baseline and after 4-10 weeks of treatment
Population: 1 patient who did not complete the treatment period due expired drug supply was not evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Gel + Oral Placebo | Placebo Gel + Oral Treatment
Number analyzed (Participants) | 12 | 14
units on a scale | 0.33 (0.64) | 0.55 (1.05)

7. Secondary Outcome: Difference in vWF Coagulation Protein in Blood Collected at Baseline and Just Prior to Surgery
Description: The difference between vWF coagulation protein in blood samples collected at baseline and before surgery were measured using the immune-turbidimetric assay.
Time Frame: Baseline to immediately before surgery (after approximately 4-10 weeks)
Population: 1 patient who did not complete the treatment period due expired drug supply was not evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percentage of vWF protein in blood
Arm/Group | Treatment Gel + Oral Placebo | Placebo Gel + Oral Treatment
Number analyzed (Participants) | 12 | 14
percentage of vWF protein in blood | -2.6 (52.3) | 51.2 (71.0)

8. Other Pre Specified Outcome: E and Z 4-OHT Isomers
Description: Descriptive statistics and confidence intervals will be provided.
Time Frame: 28-70 days
Reporting Status: Not Posted

9. Secondary Outcome: Difference in Factor VIII Coagulation Protein in Blood Collected at Baseline and Just Prior to Surgery
Description: The difference between Factor VIII coagulation protein in blood samples collected at baseline and before surgery was measured with VisuLize antigen ELISA Kits.
Time Frame: Baseline and immediately before surgery (after approximately 4-10 weeks)
Population: 1 patient who did not complete the treatment period due expired drug supply was not evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percentage Factor VIII protein in blood
Arm/Group | Treatment Gel + Oral Placebo | Placebo Gel + Oral Treatment
Number analyzed (Participants) | 12 | 14
percentage Factor VIII protein in blood | 8.7 (18.5) | 11.6 (17.3)

10. Secondary Outcome: Difference in Factor IX Coagulation Protein in Blood Collected at Baseline and Just Prior to Surgery
Description: The difference between Factor IX coagulation protein in blood samples collected at baseline and before surgery was measured with VisuLize antigen ELISA Kits.
Time Frame: Baseline and immediately before surgery (after approximately 4-10 weeks)
Population: 1 patient who did not complete the treatment period due expired drug supply was not evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percentage of Factor IX protein in blood
Arm/Group | Treatment Gel + Oral Placebo | Placebo Gel + Oral Treatment
Number analyzed (Participants) | 12 | 14
percentage of Factor IX protein in blood | -5.6 (13.6) | 0.4 (10.2)

11. Secondary Outcome: Difference in Protein S Coagulation Protein in Blood Collected at Baseline and Just Prior to Surgery
Description: The difference between protein S coagulation protein in blood samples collected at baseline and before surgery was measured using an ELISA Kit.
Time Frame: Baseline and immediately before surgery (after approximately 4-10 weeks)
Population: 1 patient who did not complete the treatment period due expired drug supply was not evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percentage of protein S in blood
Arm/Group | Treatment Gel + Oral Placebo | Placebo Gel + Oral Treatment
Number analyzed (Participants) | 12 | 14
percentage of protein S in blood | -1.6 (6.5) | -2.7 (9.3)

ADVERSE EVENTS:
Time Frame: 14 weeks
Description: Patients were asked about any adverse events they may have experienced at every study visit.
Arm/Group | Treatment Gel + Oral Placebo | Placebo Gel + Oral Treatment
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/14
Other Adverse Events (participants affected / at risk) | 12/12 | 14/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Gel + Oral Placebo (N=12) | Placebo Gel + Oral Treatment (N=14)
Sweating (Diaphoresis) (Blood and lymphatic system disorders) | 4 (10) | 6 (30)
Edema (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Hemorrhage, Gu::Vagina (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypertension (Cardiac disorders) | 0 (0) | 1 (1)
Insomnia (Endocrine disorders) | 3 | 1 (1)
Fatigue (Endocrine disorders) | 4 (4) | 5 (6)
Hot Flashes (Endocrine disorders) | 7 (13) | 7 (26)
Vision-blurred vision (Eye disorders) | 0 (0) | 1 (2)
Anorexia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 3 (3)
Heartburn/Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (5)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 5 (5) | 0 (0)
Flu -like Syndromes (General disorders) | 1 (1) | 0 (0)
Pain: Other (General disorders) | 0 (0) | 2 (2)
Pain: Back (General disorders) | 0 (0) | 1 (1)
Pain: Chest/Thorax Nos (General disorders) | 0 (0) | 1 (1)
Pain: Extremity/Limb (General disorders) | 0 (0) | 2 (4)
Pain: Headache (General disorders) | 0 (0) | 6 (8)
Pain: Pain: Nos (General disorders) | 0 (0) | 1 (1)
Pain: Pain: Stomach (General disorders) | 0 (0) | 1 (1)
Pain: Throat/Pharynx/Larynx (General disorders) | 0 (0) | 3 (3)
Fever (Immune system disorders) | 0 (0) | 1 (1)
Infection- Other (Infections and infestations) | 0 (0) | 3 (3)
Infection with unknown ANC (Infections and infestations) | 2 (2) | 1 (1)
Weight Gain (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Mood Alteration (Nervous system disorders) | 1 (1) | 3 (3)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3)
Cognitive Disturbance (Nervous system disorders) | 1 (1) | 1 (1)
Memory Impairment (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Incontinence (Renal and urinary disorders) | 0 (0) | 3 (3)
Vaginitis (not due to infection) (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal discharge (not infectious) (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Sexual/Reproductive Function - Other (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Irregular Menses (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pain: Breast (Reproductive system and breast disorders) | 5 (7) | 9 (12)
Pain: Vagina (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal Dryness (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Nasal Cavity/Paranasal Sinus Reactions (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4)
Voice change/dysarthria (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnea (shorntess of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (6)
Pain: Chest Wall (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Nail changes (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Wound complication, non-infectious (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus/Itching (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was originally designed to enroll 112 participants, unfortunately, the shelf-life of the study drug expired which resulted in early closure of the study after only 31 participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes